CLINICAL TRIAL: NCT01504152
Title: Survey to Assess International Travel Patterns and Health Preparations of Hematopoietic Stem Cell Transplant Recipients at Memorial Sloan-Kettering Cancer Center
Brief Title: International Travel Patterns and Health Preparations of Hematopoietic Stem Cell Transplant Recipients at Memorial Sloan-Kettering Cancer Center
Status: Completed | Type: Observational
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: Weill Medical College of Cornell University (Other)
Responsible Party: Sponsor
Other Study IDs: 11-176
Record Dates: First submitted 2012-01-03; First posted 2012-01-05 (Estimated); Last update posted 2013-07-12 (Estimated); Status verified 2013-07

CONDITIONS: Hematopoietic Stem Cell Transplant
Keywords: International travel; cancer patients; HSCT; Quality of Life; questionnaire; 11-176
MeSH Terms: interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective

GROUPS / COHORTS (1):
- patients who received HSCT at MSKCC between 2005-2010: A self-administered patient questionnaire will be used to collect data that will assess the prevalence of international travel after HSCT and travel related morbidity and exposure risks among HSCT recipients.
  Interventions: Behavioral: questionnaire

INTERVENTIONS:
Behavioral: questionnaire — The intervention is a self-administered questionnaire that is voluntarily completed by the subject. This questionnaire has been previously validated and demonstrated to be reproducible in English speaking travelers. The final version of the survey questionnaire consists of 49 questions.Patients who never traveled after HSCT will answer only eighteen questions related to their medical and HSCT history in addition to their demographics.

SUMMARY:
The purpose of this study is to survey patients who underwent hematopoietic stem cell transplant (HSCT) to assess if they have traveled or not internationally after transplant. This information will help to improve the understanding of the needs for travel health strategies and interventions to provide healthy and safe travel to HSCT patients. The findings of this survey will also be used to develop travel health related interventions for patients living with cancer as well.

ELIGIBILITY:
Inclusion Criteria:

* Hematopoietic Stem Cell Transplant (HSCT) recipients at MSKCC from 1/1/2005 to 12/31/2010.
* Age at HSCT ≥ 18 years
* Permanent mailing address in the United States of America

Exclusion Criteria:

* Subject unable to fill the questionnaire due to language barriers.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who received HSCT at MSKCC between 2005-2010 and were alive after the first year after HSCT.
Sampling Method: Non-Probability Sample
Enrollment: 519 (Actual)
Dates: Start 2011-12; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
prevalence of international travel | 2 years
  of the targeted patients Proportion of Hematopoietic Stem Cell Transplant (HSCT) patients who traveled internationally within two years after HSCT

SECONDARY OUTCOMES:
international travel was during a high-risk specific period | 2 years
  Proportion of patients traveling to destinations that are at high risk areas for infections
patients that sought pre-travel health advice | 2 years
  among those who traveled to high risk areas for infections
travelers that becomes ill and required medical attention | 2 years
  during or after return from international travel.

CONTACTS AND LOCATIONS:
Overall Officials: Monika Shah, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan-Kettering Cancer Center, New York, New York, United States

REFERENCES:
- See also: Memorial Sloan-Kettering Cancer Center — http://www.mskcc.org/